CLINICAL TRIAL: NCT04840654
Title: Pudendal vs Caudal Block for Pediatric Penile Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding and change of PI
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB20-1857
Record Dates: First submitted 2021-04-06; First posted 2021-04-12 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain
Keywords: Nerve Block; Caudal Block; Pudendal Block; Circumcision; Hypospadias; Postoperative Analgesia; Opioid Consumption; Pain Score
MeSH Terms: conditions — Pain, Postoperative; Hypospadias

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to 2 groups. One group will receive the Caudal block. The other group will receive the Pudendal block.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be an observer-blinded RCT. The surgeon, regional pediatric anesthesiologist, and operating room staff (anesthesiologists and nurses) will not be blinded to the treatment group. However, the patient and family, recovery room nurses, and study coordinator who collects the data from families will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Caudal block (Active Comparator): This group will receive the Caudal block during their operation (50 patients circumcision, 50 patients hypospadias). This group consist of 100 subjects
  Interventions: Procedure: Caudal Block
- Pudendal Block (Active Comparator): This group will receive the Pudendal block during their operation (50 patients circumcision, 50 patients hypospadias). This group consist of 100 subjects
  Interventions: Procedure: Pudendal Block

INTERVENTIONS:
Procedure: Caudal Block — A caudal block is a procedure that will help lessen a child's pain after an operation.
  100 subjects will be randomized to this block procedure.
  Arms: Caudal block
Procedure: Pudendal Block — form of local anesthesia commonly used in the practice of obstetrics to relieve pain during the delivery of baby by forceps.
  100 Subjects will be randomized to this block procedure.
  Arms: Pudendal Block

SUMMARY:
The study will compare recovery profile in children receiving pudendal blocks vs caudal analgesia for ambulatory circumcision or hypospadias repair in children between 6 months and 2 years. The subjects of the study will be randomized to receive either a caudal or a pudendal block.

DETAILED DESCRIPTION:
The study participation will begin on the day of surgery and end at the time of last surgical follow-up visit, approximately two weeks later. All procedure related, follow-up clinic visit and PACU data will be collected by the research team from the patient's EPIC record (demographic data, pain scores in the PACU, analgesic consumption, time to perform block, time to discharge, etc). Data pertaining to the recovery of patient at home will be collected via phone call or email to the caregiver of the child. Late complications will be identified by reviewing the follow-up surgical note.

Questionnaire Administration The physical Pain journal/questionnaires

The physical Pain journal/questionnaires will be handed out to the caregiver before discharge from the Post-Anesthesia Care Unit.

The caregiver will fill out pain scores at home in the Pain Journal. The pain scores used (FLACC and PPPM) have been extensively validated. In addition, written instructions for using the pain scores to guide pain management interventions at home will be provided. Prior to discharge, caregivers will also be educated by a member of the research team on pain evaluation using the pain score and pain management algorithm.

The caregiver will be asked to answer a short questionnaire (Postoperative Parent Survey) about their child pain in the first 24 hours after discharge from the hospital. The caregiver will receive a phone call from the research team 24-48 hours after discharge to retrieve the results of the Pain Journal and Postoperative Pain Survey.

Phone Calls Approximately 24-48 hours after the child is discharged from the hospital, a member of the study team will call the caregivers/parents to retrieve the journal responses and check on the health status of the child. During this call, if there are any adverse event that may be related to the block that was performed noted, this will be documented on the AE log and a follow-up phone call will be made approximately 7 days after to verify if the event has ended or is ongoing. Upon learning about any potential related AE, the investigator will determine its severity and relationship to the study procedure and report the event per University of Chicago guidelines.

ELIGIBILITY:
Inclusion Criteria:

* - Children Aged 6 months -3 years
* Scheduled for elective outpatient circumcision or hypospadias repair

Exclusion Criteria:

* ASA classification ≥ 3
* emergency surgery
* history of a complex regional pain syndrome
* sacral dimple
* known vertebral spinal abnormalities, spinal dysraphism
* history of long-term analgesic use
* use of any analgesic (e.g., an opioid medication, acetaminophen, or a nonsteroidal anti-inflammatory agent) within 24 hours before surgery
* history of renal insufficiency or a bleeding disorder
* concurrent additional surgery at another anatomic site
* being a ward of the state
* a non-English speaking patient or primary caregiver
* inability of the primary caregiver to comply with home instructions

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Analgesic Consumption | 24 Hours
  Number of doses of analgesics in the recovery room and in the first 24 hours at home

SECONDARY OUTCOMES:
Postoperative Pain Scores | 2 Weeks
  Analgesia will be evaluated based on the Face, Legs, Activity, Cry, Consolability (FLACC) Scale. This scale has a maximum score of 10 and a minimum score of 0, where the higher the score, the worse outcome. FLACC scores will be recorded in the PACU by the assigned recovery room nurses.
Block failure | 2 Weeks
  Block failure (inability to place block, or block failure based on increase in HR or BP >20% in response to incision)
Intraoperative opioid consumption | During Surgery
  Intraoperative opioid consumption during surgery
Time to place the block | During Surgery
  The length of time it takes to perform the block on each subject
Time to first analgesic request at home | 2 Weeks
  Time to first analgesic request at home

CONTACTS AND LOCATIONS:
Overall Officials: Leili Khorassani, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States